CLINICAL TRIAL: NCT03393026
Title: A Multi-Center, Open-Label, Single Arm and Flexible Dose Study of the Effectiveness and Safety of Oral Use Lurasidone HCl Tablet (LATUDA®) for 40-160 mg/Day in Subjects With Schizophrenia
Brief Title: A Study of Lurasidone HCl in Subjects With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Standard Chem. & Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCPF20L01TW
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Intervention Model Description: Lurasidone 40-160 mg/day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lurasidone 40-160 mg (Experimental): Lurasidone 40-160 mg
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 40-160 mg/day for 6 weeks

SUMMARY:
The study evaluates the effectiveness and safety of Lurasidone in subjects with schizophrenia over a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female aged at 20-75 years old
2. Subjects who are diagnosed with schizophrenia based on Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria
3. CGI-S≦4 (at both screening and baseline)
4. Subject is judged by the investigator to have been clinically stable for at least 4 weeks prior to baseline and in need for a switch from their current antipsychotic treatment due to insufficient clinical response or poor tolerability (side effects, metabolic complications, etc.).
5. If the subject recruits from OPD, the subject should be intolerant to the AE or is insufficient in current antipsychotics treatment by investigator's judgment.
6. Childbearing potential women who consented to the consistent use of the acceptable contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
7. Subject is able and agrees to remain off (or stable dosage) prior antipsychotic medication during the study period as defined by this protocol.
8. In the Investigator's opinion, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the investigator and to participate in, and to comply with, the requirements of the entire protocol.
9. Subject is willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject has clinically substantial risk of suicide or violent behavior as judged by the investigator.
2. Subject with the past history of neuroleptic malignant syndrome, water intoxication, paralytic ileus or dementia related psychosis
3. Subjects is active pregnancy (must have a negative pregnancy test at screening) or nursing (must not be lactating).
4. Subject has received treatment with MAO inhibitors within 14 days prior to the screening (Visit 1).
5. Subject is currently participating, or has participated in, a study with an investigational or marketed compound or device within 1 month prior to signing the informed consent.
6. Subject is unstable or critical untreated medical illness by the judgment of investigators.
7. Subject who is otherwise considered ineligible for the study by investigator. For example, subjects experienced serious medical condition including known clinically relevant laboratory abnormalities, and hypersensitivity to Lurasidone.
8. Subjects who were considered resistance to treatment for psychotic symptoms by the investigator.
9. Total daily dose of pre-switch antipsychotic was exceeded the equivalent of haloperidol 12 mg/day.
10. Subjects have received long depot neuroleptics within 4 weeks prior to enrollment. Or, subject was treated with clozapine for refractory psychosis within 1 month of enrollment.
11. Subject requires treatment with any potent CYP3A4 inhibitors or inducers during the study. Subject requires treatment with a drug that consistently prolongs the QTc interval.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
time to treatment failure. | 6 weeks
  Treatment failure is defined as any occurrence of: Insufficient clinical response Exacerbation of underlying disease Discontinuation due to adverse event

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale(PANSS) total scores | 6 weeks
  " Mean Change from baseline at week 6" in Positive and Negative Syndrome Scale total scores.
  The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item.The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity
Clinical Global Impression-Improvement (CGI-I) Scale | 6 weeks
  " Mean Change from baseline at week 6" in Clinical Global Impression-Improvement.
  The CGI-I Score is a clinician-rated assessment of the subject's overall clinical condition. The CGI-I score obtained at the baseline (initiation) visit serves as a good basis for making this assessment. This subject's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Clinical Global Impression-Severity (CGI-S) | 6 weeks
  " Mean Change from baseline at week 6" in Clinical Global Impression-Severity.
  The CGI-S Score is a clinician-rated assessment of the subject's current illness state on a 7-point scale (1-7), where a higher score is associated with greater illness severity. Following a clinical interview, the CGI-S can be completed in 1-2 minutes.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei City Hospital, Songde Branch, Taipei
  - Tri-Service General Hospital, Taipei